CLINICAL TRIAL: NCT05700617
Title: Myocardial Reserve in Advanced Heart Failure Patients
Brief Title: Cardiac Power Output in Cardiogenic Shock Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0817
Record Dates: First submitted 2022-11-01; First posted 2023-01-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Cardiogenic Shock
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic | interventions — Milrinone

STUDY DESIGN:
Intervention Model Description: prospective, observational, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1:1 Randomization to Milrinone (Active Comparator): Milrinone will be given as a bolus dose of 50 mcg/kg. If a maintenance milrinone infusion is felt to be necessary, it will be maintained at 0.125-0.375 mcg/kg/min.
  Interventions: Drug: 1:1 Randomization to receive milrinone
- 1:1 No Intervention (No Intervention): Subjects without evidence of cardiogenic shock will not receive Milrinone.

INTERVENTIONS:
Drug: 1:1 Randomization to receive milrinone — Randomized to receive either inotropic agent: milrinone or no agent
  Other Names: Milrinone
  Arms: 1:1 Randomization to Milrinone

SUMMARY:
The main purpose of this study is to determine whether differences in myocardial reserve predict clinical outcomes for heart failure patients.

DETAILED DESCRIPTION:
This study is designed as a prospective, observational, crossover study to assess the feasibility of using differences in invasive hemodynamics of cardiac function, representing myocardial reserve, to predict clinical outcomes for heart failure patients. Patients with heart failure referred for right heart catheterization (RHC) by the advanced heart failure team as part of 1) evaluation for advanced heart failure therapies, including left ventricular assist device (LVAD), orthotopic heart transplant (OHT), temporary or long-term inotrope therapy, or counter-pulsation (temporary intra-aortic balloon pump (IABP) or long-term with NuPulse device), 2) for accurate assessment of invasive hemodynamics due to worsening clinical status, 3) assessment of myocardial recovery for consideration of LVAD or NuPulse decommissioning or removal or mechanical circulatory support removal, or 4) accurate assessment of cardiac function in patients with reduced LVEF prior to valve replacement for aortic insufficiency (AI) or mitral regurgitation (MR).

ELIGIBILITY:
Inclusion Criteria:

1. LVEF ≤ 40%
2. Referred for RHC for:

   1. Evaluation for advanced heart failure therapies, including LVAD, OHT, temporary or long-term inotrope therapy, or counter-pulsation (temporary or long-term with NuPulse device OR
   2. Accurate assessment of invasive hemodynamics due to worsening clinical status, OR
   3. Assessment of myocardial recovery for consideration of LVAD or counter-pulsation (temporary IABP or long-term with NuPulse device) decommissioning or removal OR
   4. Assessment of cardiac function and valvular abnormalities prior to planned valvular surgery for MR or AI
3. Estimated glomerular filtration rate (eGFR) ≥ 30 ml/min/1.73 m2
4. Age ≥ 18 years-old
5. Intent for admission based on RHC data

Exclusion Criteria:

1. eGFR < 30 ml/min/1.73 m2
2. Severe, non-revascularized coronary artery disease
3. Concurrent acute coronary syndrome
4. Age < 18 years-old
5. History of significant ventricular arrhythmia without an ICD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in invasive hemodynamics using a pulmonary artery (PA) catheter measuring mmHg | Baseline and 6,12,24,36,72 Hours post-inotrope challenge.
  Changes invasive hemodynamics representing myocardial reserve will be measured in 5 patients using a pulmonary artery (PA) catheter:
  Pulmonary capillary wedge pressure (PCWP mmHg); Right Atrial pressure (RA mmHg); Pulmonary Atrial pressures (PA mmHg);
Changes in invasive hemodynamics using a pulmonary artery (PA) catheter measuring L/min/m2 | Baseline and 6,12,24,36,72 Hours post-inotrope challenge.
  Changes invasive hemodynamics representing myocardial reserve will be measured in 5 patients using a pulmonary artery (PA) catheter:
  Cardiac output by Fick (CO L/min/m2); Cardiac index by Fick (CI L/min/m2).
Advanced heart failure therapy | 2 years
  Duration of time without need for definitive advanced heart failure therapy (LVAD, OHT) or death.
Inotropes | 2 years
  Duration of time on inotropes during hospitalization
Death | 2 years
  Cardiovascular death and/or all-cause mortality
Cardiac output measurement using a pulmonary artery (PA) catheter measuring mmHg at 2 years | 2 years
  Efficacy of increasing cardiac output with milrinone compared to dobutamine using changes invasive hemodynamics in 5 patients using a pulmonary artery (PA) catheter:
  Pulmonary capillary wedge pressure (PCWP mmHg), Right Atrial pressure (RA mmHg), Pulmonary Atrial pressures (PA mmHg),
Cardiac output measurement using a pulmonary artery (PA) catheter measuring CO L/min/m2 at 2 years | 2 years
  Efficacy of increasing cardiac output with milrinone compared to dobutamine using changes invasive hemodynamics in 5 patients using a pulmonary artery (PA) catheter:
  Cardiac output by Fick (CO L/min/m2), Cardiac index by Fick (CI L/min/m2.)

SECONDARY OUTCOMES:
Durable support | 6 hours
  Duration of time successfully off of counterpulsation, LVAD, or ECMO support
Durable support | 12 hours
  Duration of time successfully off of counterpulsation, LVAD, or ECMO support
Durable support | 24 hours
  Duration of time successfully off of counterpulsation, LVAD, or ECMO support
Durable support | 36 hours
  Duration of time successfully off of counterpulsation, LVAD, or ECMO support
Durable support | 48 hours
  Duration of time successfully off of counterpulsation, LVAD, or ECMO support
Durable support | 72 hours
  Duration of time successfully off of counterpulsation, LVAD, or ECMO support
Hospital discharge | Up to 12 weeks
  Hospital discharge without LVAD, OHT, home-inotropes, long-term counter-pulsation device (i.e NuPulse), or death.
  Patients will be monitored at the the following timepoints while admitted in the Cardiac Intensive Care Unit (CICU) 12 Hours 24 Hours 36 Hours 48 Hours 72 Hours
Home inotropic | 2 years
  Duration of time on home inotropic agents
LVAD decommissioning measuring mmHg | 2 years
  If a patient is enrolled in the study that has an left ventricular assist device (LVAD) decommissioning or removal (not due to open heart transplant, pump malfunction, or death) the following will be assessed:
  A. Changes in invasive hemodynamics using a pulmonary artery (PA) catheter:
  Pulmonary capillary wedge pressure (PCWP mmHg) Right Atrial pressure (RA mmHg) Pulmonary Atrial pressures (PA mmHg)
LVAD decommissioning measuring L/min/m2 | 2 years
  If a patient is enrolled in the study that has an left ventricular assist device (LVAD) decommissioning or removal (not due to open heart transplant, pump malfunction, or death) the following will be assessed:
  A. Changes in invasive hemodynamics using a pulmonary artery (PA) catheter:
  1. Cardiac output by Fick (CO L/min/m2)
  2. Cardiac index by Fick (CI L/min/m2)
  B. Myocardial reserve (i.e. cardiac power output, aortic pulsatility index, Cardiac output by Fick (CO L/min/m2) Cardiac index by Fick (CI L/min/m2)) after inotrope challenge.
  C. Association of myocardial reserve with other known variables of cardiovascular and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Valluvan Jeevanandam, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu S, Thiruvengadam SK, Sciortino CM, Russell SD, Schulman SP. Predictors of intra-aortic balloon pump hemodynamic failure in non-acute myocardial infarction cardiogenic shock. Am Heart J. 2018 May;199:181-191. doi: 10.1016/j.ahj.2017.11.016. Epub 2017 Dec 13. PMID 29754660
- [Background] Zhang X, Wang Z, Zhang L, Zhao X, Han Y. Comparative Effectiveness and Safety of Intermittent, Repeated, or Continuous Use of Levosimendan, Milrinone, or Dobutamine in Patients With Advanced Heart Failure: A Network and Single-Arm Meta-analysis. J Cardiovasc Pharmacol. 2024 Jul 1;84(1):92-100. doi: 10.1097/FJC.0000000000001561. PMID 38547524
- [Background] Gayatri D, Tongers J, Efremov L, Mikolajczyk R, Sedding D, Schumann J. Prophylactic use of inotropic agents for the prevention of low cardiac output syndrome and mortality in adults undergoing cardiac surgery. Cochrane Database Syst Rev. 2024 Nov 27;11(11):CD013781. doi: 10.1002/14651858.CD013781.pub2. PMID 39601298
- [Result] Fincke R, Hochman JS, Lowe AM, Menon V, Slater JN, Webb JG, LeJemtel TH, Cotter G; SHOCK Investigators. Cardiac power is the strongest hemodynamic correlate of mortality in cardiogenic shock: a report from the SHOCK trial registry. J Am Coll Cardiol. 2004 Jul 21;44(2):340-8. doi: 10.1016/j.jacc.2004.03.060. PMID 15261929